CLINICAL TRIAL: NCT01266083
Title: Phase 2 Trial of a WT1 Analog Peptide Vaccine in Patients in Complete Remission (CR) From Acute Myeloid Leukemia (AML) or Acute Lymphoblastic Leukemia (ALL)
Brief Title: WT1 Vaccine Treatment of Patients in Remission From Acute Myeloid Leukemia (AML) or Acute Lymphoblastic Leukemia (ALL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sellas Life Sciences Group (Industry)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-143
Expanded Access: NCT05593185 (Available)
Record Dates: First submitted 2010-12-21; First posted 2010-12-24 (Estimated); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia
Keywords: Galinpepimut-S; WT1 analog peptide vaccine; 10-143; Wilms Tumor-1 protein; SLS-001; complete remission; overall survival
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Pathologic Complete Response | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Monatide (IMS 3015)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Galinpepimut-S + Montanide + GM-CSF (Experimental): Galinpepimut-S (GPS) and Montanide (in a 1 mL emulsion) are administered subcutaneously (s.c.) Q2W on weeks 0, 2, 4, 6, 8, and 10. GM-CSF (70 μg) are administered s.c. one to two days before and on the day of GPS/Montanide administration. Participants with no recurrence after Week 12 and who are clinically stable may be eligible to receive up to 6 additional monthly vaccinations.
  Interventions: Biological: Galinpepimut-S; Biological: GM-CSF; Other: Montanide

INTERVENTIONS:
Biological: Galinpepimut-S — Galinpepimut-S admixed with the adjuvant Montanide following specified schedule
  Other Names: GPS; SLS-001
Biological: GM-CSF — subcutaneous injection
  Other Names: sargramostim
Other: Montanide — adjuvant

SUMMARY:
This trial will assess the safety and efficacy of vaccination with galinpepimut-S (GPS), a WT1 peptide vaccine, in patients who are in complete remission from leukemia.

Participants will receive vaccinations with GPS every 2 weeks for 10 weeks (a total of 6 vaccinations). In the absence of disease recurrence at Week 12 and if clinically stable after the first 6 vaccinations, participants may continue to receive up to six more vaccinations every month.

DETAILED DESCRIPTION:
This clinical study is conducted in patients in complete remission from acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL). The primary objective is to assess the effect of vaccination with galinpepimut-S (GPS) on patient survival and the safety profile.

Galinpepimut-S (GPS) consists of four WT1-derived peptides which have been chosen to strengthen antigenicity, but also broaden immunogenicity over a wide range of HLA subtypes, being able to stimulate both CD8+ (MHC Class I)- and CD4+ (MHC Class II)-dependent responses. Galinpepimut-S is administered with the adjuvant Montanide and sargramostim (GM-CSF).

Participants will receive vaccinations with GPS every 2 weeks for 10 weeks (a total of 6 vaccinations). In the absence of disease recurrence at Week 12 evaluation and if clinically stable after the first 6 vaccinations, participants may continue to receive up to six more vaccinations every month. Following the last vaccination, participants will be followed regularly (every 1 to 3 months) in an outpatinet setting for up to 3 years from the first treatment date.

ELIGIBILITY:
Inclusion Criteria:

* Morphologic confirmation of a diagnosis of AML or ALL at MSKCC
* Patients will have completed induction therapy, achieved 1st CR and will have completed any planned postremission therapy. Patients are not candidates for allogeneic stem cell transplantation. For purposes of this study, patients who are not candidates for allogeneic stem cell transplantation shall be defined as 1) those who do not meet the eligibility criteria of an open allogeneic transplant protocol or 2) those who do not have a suitable available HLA matched donor available or 3) those who refuse to undergo stem cell transplantation or 4) those patients whose disease is characterized by "good risk" features (For AML the following cytogenetic subtypes: t(8;21), inv (16), or t(16;16), t(15;17), normal karyotype with mutated NPM1 and negative for tandem duplication of FLT-3. For ALL: T cell phenotype of any B lineage disease exclusive of t(9;22) or t(4;11) in whom allogenic stem cell transplantation in 1st CR would not be offered as standard of care.
* Alternatively, those patients greater than or equal to 60 years of age who have achieved 1st CR and in whom no further postremission chemotherapy is planned may be enrolled
* Patients must have documented WT1 + disease. For purpose of this study, this is defined as detectable presence of any WT1 transcript via RT-PCR on a bone marrow performed at MSKCC within 4 weeks prior to the administration of the first dose of vaccine.
* Patients must be within 2 years of achieving CR following chemotherapy
* At least 4 weeks must have elapsed between the patient's last chemotherapy or radiation treatment and the first vaccination.
* Age ≥ 18 years
* Karnofsky performance status ≥ 50%
* Hematologic parameters:

Absolute neutrophil count (ANC) ≥ 1000/μL

* Platelets > 50 k/μL

Biochemical parameters:

* Total bilirubin ≤ 2.0 mg/dL AST and ALT ≤ 2.5 x upper limits of normal
* Creatinine ≤ 2.0 mg/dL

Exclusion Criteria:

* Pregnant or lactating women
* Patients with documented evidence of leptomeningeal disease
* Patients who have undergone autologous or allogeneic stem cell transplantation
* Patients with active infection requiring systemic antimicrobials
* Patients taking systemic corticosteroids
* Patients with serious unstable medical illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-01-14 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Maslak, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maslak PG, Dao T, Bernal Y, Chanel SM, Zhang R, Frattini M, Rosenblat T, Jurcic JG, Brentjens RJ, Arcila ME, Rampal R, Park JH, Douer D, Katz L, Sarlis N, Tallman MS, Scheinberg DA. Phase 2 trial of a multivalent WT1 peptide vaccine (galinpepimut-S) in acute myeloid leukemia. Blood Adv. 2018 Feb 13;2(3):224-234. doi: 10.1182/bloodadvances.2017014175. PMID 29386195
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Galinpepimut-S + Montanide + GM-CSF
Started | 22
Eligible for Additional Monthly Vaccinations After Initial 6 Vaccinations (Q2W) | 13
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Galinpepimut-S + Montanide + GM-CSF
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 64 [25 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 7
Karnofsky performance status [Mean (Standard Deviation); unit: scores on a scale] — Karnofsky Performance Scale (KPS) Index classifies the patient's functional impairment and assesses individual patient's prognosis. Although the total range is 0-100, the minimum score eligible to enter the study is 50 or greater.
  Low KPS scores equate to worse prognosis. 80 to 100: Able to carry on normal activity; no special care needed. 50 to 70: Cares for self; unable to carry on normal activity; varying amount of assistance needed.
  0-40: (ineligible to enter study) Unable to care for self; requires equivalent of institutional or hospital care; disease may be progressing rapidly.
  scores on a scale | 93.8 (5.9)
HLA-A* 02:01 positive [Count of Participants; unit: Participants] | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: OS at 3 years, measured from first treatment with GPS to patient's survival status at 3 years or more
Time Frame: 3 years
Population: Of the 22 patients, 19 (86.4%) were evaluable for survival at 3 years,
Measure: Number; unit: percentage of participants
Arm/Group | Galinpepimut-S + Montanide + GM-CSF
Number analyzed (Participants) | 19
percentage of participants | 47

2. Secondary Outcome: Progression-free Survival
Description: Time to PFS measured from first administration of GPS to relapse or death from any cause
Time Frame: 5 years and 8 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Galinpepimut-S + Montanide + GM-CSF
Number analyzed (Participants) | 22
days | 283 [71 to NA] — Upper limit of the 95% confidence interval was not reached at 5 years and 8 months due to end of study monitoring

ADVERSE EVENTS:
Time Frame: 5 years, 8 months
Arm/Group | Galinpepimut-S + Montanide + GM-CSF
All-Cause Mortality (participants affected / at risk) | 10/22
Serious Adverse Events (participants affected / at risk) | 1/22
Other Adverse Events (participants affected / at risk) | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galinpepimut-S + Montanide + GM-CSF (N=22)
Non-cardiac chest pain (Cardiac disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Galinpepimut-S + Montanide + GM-CSF (N=22)
Injection Site Reaction (General disorders) | 10
Skin Induration (Skin and subcutaneous tissue disorders) | 7
Fatigue (General disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 6
Lymphocyte Count Decreased (Investigations) | 6
Neutrophil Count Decreased (Investigations) | 6
White Blood Cell Count Decreased (Investigations) | 6
Platelet Count Decreased (Investigations) | 4
Pain (General disorders) | 3
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3
Flushing (Vascular disorders) | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2
Skin Infection (Infections and infestations) | 2
Upper Respiratory Tract Infection (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 2
Headache (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes